CLINICAL TRIAL: NCT00738179
Title: Sleep Apnea cardioVascular Endpoints Study - Investigating the Effectiveness of Treatment With CPAP vs Standard Care in Reducing CV Morbidity and Mortality in Patients With Co-existing CV Disease and Moderate-severe Obstructive Sleep Apnea.
Brief Title: Continuous Positive Airway Pressure Treatment of Obstructive Sleep Apnea to Prevent Cardiovascular Disease
Acronym: SAVE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adelaide Institute for Sleep Health (Other)
Collaborators: Philips Respironics (Industry); National Health and Medical Research Council, Australia (Other); ResMed (Industry); Fisher and Paykel Healthcare (Industry); The George Institute (Other); Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Professor R. Doug McEvoy, MD, Director, Adelaide Institute for Sleep Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAVE001; ANZCTR 12608000409370
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Sleep Apnea; Cardiovascular Disease
Keywords: Continuous Positive Airway Pressure (CPAP); Obstructive Sleep Apnea (OSA); Cardiovascular (CV); Cardiovascular Disease; Clinical Trial
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CPAP plus standard care of cardiovascular risk factors
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- 2 (Active Comparator): Standard care alone
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — CPAP worn nightly
  Arms: 1
Other: Standard care — Standard care of cardiovascular risk factors
  Arms: 2

SUMMARY:
Obstructive Sleep Apnea (OSA) is a condition in which a person stops breathing for several seconds at a time due to relaxation of the throat muscles. This can occur many times during sleep. It is known to cause sleepiness and poor concentration during the day. Research indicates that OSA may be a modifiable risk factor for cardiovascular disease due to its association with hypertension, stroke, heart attack and sudden death. The standard therapy for symptomatic OSA is continuous positive airway pressure (CPAP). CPAP has been shown to effectively reduce snoring, obstructive episodes and daytime sleepiness and to modestly reduce blood pressure and other risk factors for cardiovascular disease. The overall aim of SAVE is to determine if CPAP can reduce the risk of heart attack, stroke or heart failure for people with OSA.

DETAILED DESCRIPTION:
There is increasing evidence to indicate that OSA is an important modifiable risk factor for CV disease including stroke, MI, and heart failure. Increased nocturnal arterial blood pressure (BP), hypercoagulability, oxidative stress, inflammation, insulin resistance and cardiac arrhythmias are all associated with OSA. These effects are presumed to accelerate the progression of atheromatous disease, particularly within the coronary or cerebral vasculature. Moreover, OSA also appears to increase the risk of sudden death during sleep, which is different from the circadian pattern of sudden death in those without OSA, suggesting that episodes of apnea may have a direct triggering effect for cardiac arrhythmias or MI.

CPAP is now standard therapy for symptomatic OSA, with adherence to treatment comparable to that of other therapies for common chronic diseases. CPAP can eliminate apneas and improve daytime sleepiness, mood and quality of life. Furthermore, short term (1-3 months) randomised controlled trials of CPAP have shown modest reductions in blood pressure (BP) and other markers of CV disease, including C-reactive protein (CRP) and coagulation. However, the epidemiological data is complicated by potential residual confounding factors and the randomised evidence is limited. Thus, a direct causal link between OSA and CV disease remains inconclusive. The management of OSA, therefore, remains principally directed towards symptom control rather than CV risk modification.

The present trial aims to test whether long-term use of CPAP can reduce the incidence of CV events. If the trial shows that CPAP treatment of OSA reduces the incidence of CV events it will influence clinical practice toward the early detection and management of OSA, and add CPAP to the range of strategies available for the prevention of CV disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, any race, and aged between 45 and 75 years
2. Evidence of established coronary or cerebrovascular disease as evident by:

   * Coronary artery disease

     * Previous MI (equal to or greater than 90 days prior to ApneaLinkTM assessment)
     * Stable angina or unstable angina (Clinical event equal to or greater than 30 days and confirmatory test equal to or greater than 7 days prior to ApneaLinkTM assessment) defined as either ≥70% diameter stenosis of at least one major epicardial artery segment, or ≥50% diameter stenosis of the left main coronary artery, or >50% stenosis in at least two major epicardial arteries.; or positive stress test (ST depression equal to or greater than 2 mm or a positive nuclear perfusion scintigram)
     * Multi-vessel percutaneous angioplasty (PTCA) and/or stent equal to or greater than 90 days prior to ApneaLinkTM assessment
     * Multi-vessel coronary artery bypass surgery (CABG) >1 year prior to ApneaLinkTM assessment
   * Cerebrovascular disease

     * Previous stroke (includes definite or presumed cerebral ischaemia/infarction and intracerebral but not subarachnoid haemorrhage) equal to or greater than 90 days prior to ApneaLinkTM assessment or minor disabling stroke with minimal residual neurological disability (modified Rankin Score of '0 = no symptoms' or '1 = No significant disability despite symptoms, able to carry out all usual duties and activities' within 7 days of stroke onset) ≥7 days prior to ApneaLinkTM assessment.
     * Previous transient ischaemic event (TIA) of the brain or retina (symptoms <24 hours) but not of presumed vertebrobasilar system ischemia. The TIA diagnosis must be confirmed by a suitably qualified clinician (≥7 days but <1year prior to ApneaLinkTM assessment)
3. Patients have moderate-severe OSA (equivalent to apnea plus hypopneas index [AHI] >30 per hour of sleep) as determined by a ≥ 4% oxygen dip rate > 12/ h on overnight testing using the ApneaLinkTM device and confirmed by the SAVE core lab in Adelaide upon receipt of the ApneaLinkTM data
4. Patients are able and willing to give appropriate informed consent

Exclusion Criteria:

Patients will be excluded from entry if ANY of the criteria listed below are met:

1. Any condition that in the opinion of the responsible physician or investigator makes the potential participant unsuitable for the study. For example,

   * co-morbid disease with severe disability or likelihood of death
   * significant memory, perceptual, or behavioural disorder
   * neurological deficit (e.g. limb paresis) preventing self administration of the CPAP mask
   * contraindication to CPAP use e.g. pneumothorax
   * residence sufficiently remote from the clinic to preclude follow-up clinic visits
2. Any planned coronary or carotid revascularisation procedure in the next 6 months
3. Severe respiratory disease defined as

   * severe chronic obstructive pulmonary disease (FEV1/FVC < 70% and FEV1 < 50% predicted), or
   * resting, awake SaO2 < 90% by ApneaLinkTM device
4. New York Heart Association (NYHA) categories III-IV of heart failure
5. Other household member enrolled in SAVE trial or using CPAP
6. Prior use of CPAP treatment for OSA
7. Increased risk of a sleep-related accident and/or excessive daytime sleepiness, defined by any one of the following:

   * driver occupation (eg truck, taxi)
   * 'fall-asleep' accident or 'near miss' accident in previous 12 months
   * high (> 15) score on the Epworth Sleepiness Scale
8. Severe nocturnal desaturation documented on the ApneaLinkTM device as > 10% overnight recording time with arterial oxygen saturation of < 80%
9. Cheyne-Stokes Respiration (CSResp)

   * CSResp identified on ApneaLinkTM nasal pressure recording by typical crescendo-decrescendo pattern of respiration with associated apneas and/or hypopneas in the absence of inspiratory flow limitation.
   * patients excluded if > 50% of nasal pressure - defined apneas and hypopneas judged to be due to CSResp.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2008-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
A composite of the CV endpoints of CV death, non-fatal acute myocardial infarction, non-fatal stroke, hospital admission for heart failure, and new hospitalisation for unstable angina or transient ischaemic attack. | Reviewed 6-monthly; average patient follow up, 4.5 years

SECONDARY OUTCOMES:
Composite of CV death, MI & ischaemic stroke; components of primary composite endpoint; re-vascularisation procedures; all-cause death; new onset atrial fibrillation; new onset diabetes; OSA symptom scores; mood; health-related quality of life. | Reviewed 6-monthly; average patient follow up, 4.5 years.
In a sub-sample of 600 subjects pathophysiological mechanisms of CPAP-induced CV event reduction will be explored by assessing various intermediate markers of CV risk | baseline and at 6-months, 2 and 4 years following randomisation
Cardiac MRI to assess effects of CPAP on cardiac structure and function. | Randomisation and at 6 months follow-up
  In a sub-sample of 150 participants (75 from the CPAP plus standard treatment and 75 from the standard treatment arms) the effect of CPAP on cardiac and vascular function using cardiac MRI will be investigated. The sub-study will evaluate left and right ventricular mass, volume and systolic/diastolic function and compliance of the aorta.

CONTACTS AND LOCATIONS:
Overall Officials: R D McEvoy, Principal Investigator — Adelaide Institute for Sleep Health
Locations (5):
- Adelaide Institute for Sleep Health, Repatriation General Hospital, Adelaide, South Australia, Australia
- Brazil Principal Investigator: Geraldo Lorenzi Filho, Heart Institute, University of São Paulo, São Paulo, Brazil
- Regional Coordinating Centre China: The George Institute China Beijing, Beijing, Beijing Municipality, China
- Regional Coordinating Centre India: The George Institute India 839C, Road No. 44A Jubilee Hills, Hyderabad, Andhra Pradesh, India
- Regional Coordinating Centre Spain: Spanish Respiratory Society (Sociedad Española de Neumología y Cirugía Torácica) (SEPAR), Barcelona, Spain

REFERENCES:
- [Derived] Cheng Y, Ou Q, Chen B, Loffler KA, Doug McEvoy R, Xu Y, Wang Q, Lao M. The changes of AHI after long-term CPAP in patients with comorbid OSA and cardiovascular disease. Sleep Breath. 2023 May;27(2):511-518. doi: 10.1007/s11325-022-02633-y. Epub 2022 May 14. PMID 35562555
- [Derived] Lao M, Cheng Y, Gao X, Ou Q. The interaction among OSA, CPAP, and medications in patients with comorbid OSA and cardiovascular/cerebrovascular disease: a randomized controlled trial. BMC Pulm Med. 2022 Mar 21;22(1):99. doi: 10.1186/s12890-022-01879-2. PMID 35313858
- [Derived] Stevens D, Loffler KA, Buman MP, Dunstan DW, Luo Y, Lorenzi-Filho G, Barbe FE, Anderson CS, McEvoy RD; SAVE investigators. CPAP increases physical activity in obstructive sleep apnea with cardiovascular disease. J Clin Sleep Med. 2021 Feb 1;17(2):141-148. doi: 10.5664/jcsm.8792. PMID 32951632
- [Derived] Li J, McEvoy RD, Zheng D, Loffler KA, Wang X, Redline S, Woodman RJ, Anderson CS. Self-reported Snoring Patterns Predict Stroke Events in High-Risk Patients With OSA: Post Hoc Analyses of the SAVE Study. Chest. 2020 Nov;158(5):2146-2154. doi: 10.1016/j.chest.2020.05.615. Epub 2020 Jul 15. PMID 32679238
- [Derived] Loffler KA, Heeley E, Freed R, Meng R, Bittencourt LR, Gonzaga Carvalho CC, Chen R, Hlavac M, Liu Z, Lorenzi-Filho G, Luo Y, McArdle N, Mukherjee S, Yap HS, Zhang X, Palmer LJ, Anderson CS, McEvoy RD, Drager LF; SAVE Substudy Investigators. Continuous Positive Airway Pressure Treatment, Glycemia, and Diabetes Risk in Obstructive Sleep Apnea and Comorbid Cardiovascular Disease. Diabetes Care. 2020 Aug;43(8):1859-1867. doi: 10.2337/dc19-2006. Epub 2020 Apr 14. PMID 32291275
- [Derived] Li J, Zheng D, Loffler KA, Wang X, McEvoy RD, Woodman RJ, Luo Y, Lorenzi-Filho G, Barbe F, Tripathi M, Anderson CS; SAVE Investigators. Sleep duration and risk of cardiovascular events: The SAVE study. Int J Stroke. 2020 Oct;15(8):858-865. doi: 10.1177/1747493020904913. Epub 2020 Feb 3. PMID 32013799
- [Derived] Van Ryswyk E, Anderson CS, Antic NA, Barbe F, Bittencourt L, Freed R, Heeley E, Liu Z, Loffler KA, Lorenzi-Filho G, Luo Y, Margalef MJM, McEvoy RD, Mediano O, Mukherjee S, Ou Q, Woodman R, Zhang X, Chai-Coetzer CL. Predictors of long-term adherence to continuous positive airway pressure in patients with obstructive sleep apnea and cardiovascular disease. Sleep. 2019 Oct 9;42(10):zsz152. doi: 10.1093/sleep/zsz152. PMID 31587046
- [Derived] Ou Q, Chen B, Loffler KA, Luo Y, Zhang X, Chen R, Wang Q, Drager LF, Lorenzi-Filho G, Hlavac M, McArdle N, Mukherjee S, Mediano O, Barbe F, Anderson CS, McEvoy RD, Woodman RJ; SAVE investigators. The Effects of Long-term CPAP on Weight Change in Patients With Comorbid OSA and Cardiovascular Disease: Data From the SAVE Trial. Chest. 2019 Apr;155(4):720-729. doi: 10.1016/j.chest.2018.08.1082. Epub 2018 Sep 27. PMID 30268694
- [Derived] Loffler KA, Heeley E, Freed R, Anderson CS, Brockway B, Corbett A, Chang CL, Douglas JA, Ferrier K, Graham N, Hamilton GS, Hlavac M, McArdle N, McLachlan J, Mukherjee S, Naughton MT, Thien F, Young A, Grunstein RR, Palmer LJ, Woodman RJ, Hanly PJ, McEvoy RD; SAVE (Sleep Apnea Cardiovascular Endpoints) Investigators. Effect of Obstructive Sleep Apnea Treatment on Renal Function in Patients with Cardiovascular Disease. Am J Respir Crit Care Med. 2017 Dec 1;196(11):1456-1462. doi: 10.1164/rccm.201703-0603OC. PMID 28743190
- [Derived] McEvoy RD, Antic NA, Heeley E, Luo Y, Ou Q, Zhang X, Mediano O, Chen R, Drager LF, Liu Z, Chen G, Du B, McArdle N, Mukherjee S, Tripathi M, Billot L, Li Q, Lorenzi-Filho G, Barbe F, Redline S, Wang J, Arima H, Neal B, White DP, Grunstein RR, Zhong N, Anderson CS; SAVE Investigators and Coordinators. CPAP for Prevention of Cardiovascular Events in Obstructive Sleep Apnea. N Engl J Med. 2016 Sep 8;375(10):919-31. doi: 10.1056/NEJMoa1606599. Epub 2016 Aug 28. PMID 27571048
- [Derived] Antic NA, Heeley E, Anderson CS, Luo Y, Wang J, Neal B, Grunstein R, Barbe F, Lorenzi-Filho G, Huang S, Redline S, Zhong N, McEvoy RD. The Sleep Apnea cardioVascular Endpoints (SAVE) Trial: Rationale, Ethics, Design, and Progress. Sleep. 2015 Aug 1;38(8):1247-57. doi: 10.5665/sleep.4902. PMID 25669180
- [Derived] Chai-Coetzer CL, Luo YM, Antic NA, Zhang XL, Chen BY, He QY, Heeley E, Huang SG, Anderson C, Zhong NS, McEvoy RD. Predictors of long-term adherence to continuous positive airway pressure therapy in patients with obstructive sleep apnea and cardiovascular disease in the SAVE study. Sleep. 2013 Dec 1;36(12):1929-37. doi: 10.5665/sleep.3232. PMID 24293768
- See also: Related Info — http://www.savetrial.org